CLINICAL TRIAL: NCT04556253
Title: A Multicenter, Open-Label, Phase II Study of Anti-PD-1/CTLA-4 Bispecific Antibody AK104 in the Perioperative Treatment of Locally Advanced Microsatellite Instability/Mismatch Repair Protein-Deficient Gastric and Colorectal Cancers
Brief Title: AK104 in Locally Advanced MSI-H/dMMR Gastric Carcinoma and Colorectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Jiafu Ji, Head of Beijing Cancer Hospital, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-002
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: MSI-H/dMMR Gastric Carcinoma and Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): Subjects will receive AK104 by intravenous administration.
  Interventions: Drug: AK104

INTERVENTIONS:
Drug: AK104 — Subjects will receive AK104 by intravenous administration.

SUMMARY:
This is a single-arm, multicenter phase II clinical study. The aim is to evaluate the safety, tolerability, and anti-tumor activities of AK104(a PD-1/CTLA-4 bispecific antibody) in MSI-H/dMMR locally advanced gastric adenocarcinoma and colorectal cancer during the perioperative period.Eligible patients will receive AK104 for three cycles before surgery and at most 6 months after surgery. The primary endpoint is the pathological complete response rate.

ELIGIBILITY:
Inclusion Criteria:

* Written and signed informed consent.
* Eastern Cooperative Oncology Group (ECOG) Performance Score of 0 or
* The estimated life expectancy of ≥3 months.
* Confirmed MSI-H/dMMR status by the central laboratory.
* For cohort 1, histologically or cytologically documented locally advanced gastric carcinoma(cT3-T4a, Nx, M0). For cohort 2, histologically or cytologically documented locally advanced colorectal cancer(cT2-T4a, Nx, M0).
* Haven't received any chemotherapy or radiotherapy.
* Adequate organ function.
* All female and male subjects of reproductive potential must agree to use an effective method of contraception, as determined by the Investigator, during and for 120 days after the last dose of study treatment.

Exclusion Criteria:

* Is currently participating in a study of an investigational agent or using an investigational device;
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy within 2 years prior to the first dose of study treatment;
* Has undergone major surgery within 30 days of Study Day 1;
* Has a known additional malignancy that is progressing or requires systemic treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
* Has known active central nervous system (CNS) metastases;
* Has carcinomatous meningitis;
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment NOTE: Subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study;
* Has an active infection requiring systemic therapy;
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected);
* History of myocardial infarction, unstable angina, cardiac or other vascular stenting, angioplasty, or surgery within 12 months prior to day 1 of study treatment;
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of this subject to participate, in the opinion of the treating investigator;
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study;
* Has received a live virus vaccine within 30 days of the planned first dose of study therapy;
* Is pregnant, breastfeeding, or expecting to conceive or father a child within the projected duration of the study including 120 days following the last dose of study treatment;
* Has any concurrent medical condition that, in the opinion of the Investigator, would complicate or compromise compliance with the study or the well-being of the subject.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2024-02-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
The rate of pathologic complete response(pCR%) | through study completion, an average of 1 year
  The rate of pathologic complete response evaluated by investigator

CONTACTS AND LOCATIONS:
Overall Officials: Jiafu Ji, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Peking University Cancer Hospital & Institute, Beijing, Beijing Municipality, China